CLINICAL TRIAL: NCT05164757
Title: Female Asian Nonsmoker Screening Study (FANSS)
Brief Title: Female Asian Nonsmoker Screening Study
Acronym: FANSS
Status: Active, not recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 20-00212
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serial specimens of blood will be collected at the initial screen from each subject. In addition, paraffin blocks from resected lung tumors from any subject who have any pathological specimens from the lung will be collected retrospectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study team propose to develop a database and biorepository of Asian female never smokers. This population is at increased risk for developing lung cancer but do not meet current lung cancer screening criteria. Study procedures will include up to 3 low-dose CT (LDCT) scans and a blood-based assay with the capability for early detection of cancer. Clinical, demographic and exposure history including possible WTC exposure will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-74 years
* Female
* Never Smoker defined as a lifetime exposure of less than 100 cigarettes
* Identify as from Asian descent, defined as having reported ancestry or race from the continent of Asia. Individuals with mixed heritage are eligible.

Exclusion Criteria:

* Prior history of lung cancer.
* Treatment for, or advisement by a physician of evidence of any cancer within the past five years, with the exceptions of non-melanoma skin cancer and most in-situ carcinomas based on PI discretion. (Treatment for, or evidence of, melanoma or in-situ bladder/transition cell carcinomas within the preceding five years renders the potential participant ineligible.)
* Participation in a cancer prevention trial.
* Present symptoms suggestive of current lung cancer, including: unexplained weight loss of over 15 pounds within the 12 months or unexplained hemoptysis.
* Medical or psychiatric condition precluding informed medical consent.
* Pneumonia or acute respiratory infection within 12 weeks of enrollment that was treated with antibiotics under physician supervision.

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women of Asian/Asian continent ancestry and ethnic groups are eligible for this trial.
Sampling Method: Non-Probability Sample
Enrollment: 1041 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2035-03 (Estimated); Study Completion 2035-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants who inquire about the program and are eligible to proceed with the Low Dose Computed Tomography (LDCT) screening test | Screening (Day -28 to -1)
Number of Participants who undergo initial LDCT | Visit 2 (Day 30 +/- 7)

SECONDARY OUTCOMES:
Number of diagnoses of lung cancer | Visit 2 (Day 30 +/- 7)
Number of diagnoses of lung cancer | Visit 4 (Day 365 +/- 14)
Number of diagnoses of lung cancer | Visit 6 (day 730 +/- 14)
Detection rate of Incidental thyroid nodules | Visit 2 (Day 30 +/- 7)
Detection rate of Incidental thyroid nodules | Visit 4 (Day 365 +/- 14)
Detection rate of Incidental thyroid nodules | Visit 6 (day 730 +/- 14)
Detection rate of Incidental coronary artery disease | Visit 2 (Day 30 +/- 7)
Detection rate of Incidental coronary artery disease | Visit 4 (Day 365 +/- 14)
Detection rate of Incidental coronary artery disease | Visit 6 (day 730 +/- 14)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Shum, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to FANSS@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.